CLINICAL TRIAL: NCT04821336
Title: Cholesterol Metabolites (Dendrogenin A or DDA, 6-oxo-cholestane-3β,5α-diol or OCDO,...) Quantification in Malignant Versus Normal Human Thyroid Tissue Refractory to Iodine
Brief Title: Cholesterol Metabolites Analysis in Human Thyroid and Iodine Resistance
Acronym: OXYTHYR
Status: Completed | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Cancer Research Center of Toulouse (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21HLVADS01
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-12

CONDITIONS: Thyroid Cancer
Keywords: cholesterol metabolites; dendrogenin A (DDA); 6-oxo-cholestane-3β,5α-diol (OCDO); 5,6 epoxy cholesterol; thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — frozen human thyroid samples (benign or malignant) paraffin embedded human thyroid tissue collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroid tissue samples: from 30 patients, tissue samples , frozen and embedded paraffin have been collected and preserved for research. For this study, tumoral tissue and healthy tissue will be used;
  Interventions: Other: Metabolites dosage

INTERVENTIONS:
Other: Metabolites dosage — On samples investigators will quantify cholesterol metabolite and dendrogenin A (DDA) and 6-oxo-cholestane-3β,5α-diol (ou OCDO) metabolites in malignant tissue sample on one hand, and in sane samples on other hand.
  The investigators will compare the rate of deregulation between sane and malignant ones.

SUMMARY:
The study team previously shown that a cholesterol metabolite, dendrogenin A (DDA) differentiates anaplastic thyroid cancer cell lines and that its mRNA expression is diminished in human radioiodine refractory thyroid cancer samples. The team aim to quantify via mass spectrometry and immunohistochemistry DDA and other cholesterol metabolites in thyroid cancer versus healthy thyroid tissue human samples.

DETAILED DESCRIPTION:
Retrospective study to analyze tissue samples of patients after thyroid surgery at Claudius Regaud Institute Toulouse, France, for thyroid cancer or thyroid aggressive lymphoma or benign thyroid pathology or other head&neck pathology necessitating total thyroidectomy despite normal thyroid.

Analysis focused on cholesterol metabolites quatification by mass spectrometry in liquid and gas phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone surgery at Institut Claudius Regaud for thyroid or laryngeal cancer confirmed by histology.
* Patients who have consented before surgery, for the use of participants samples for future researches.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of dendrogenin A (DDA) and 6-oxo-cholestane-3β,5α-diol (OCDO) in thyroid tissue (healthy or malignant) | 12 months after the beginning of the study
  The measurement expressed in ng / g of thyroid tissue

SECONDARY OUTCOMES:
Presence of enzymes involved in dendrogenin A (DDA) and 6-oxo-cholestane-3β,5α-diol (OCDO) production | 12 months after the beginning of the study
  intensity of signal in Liquid Chromatography-Mass Spectrometry
Number of enzymes involved in denrognenin A (DDA) and 6-oxo-cholestane-3β,5α-diol (OCDO) production | 12 months after the beginning of the study
  Quantify by immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Claudius regaud IUCT Oncopole, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Zerdoud S, Giraudet AL, Leboulleux S, Leenhardt L, Bardet S, Clerc J, Toubert ME, Al Ghuzlan A, Lamy PJ, Bournaud C, Keller I, Sebag F, Garrel R, Mirallie E, Groussin L, Hindie E, Taieb D. Radioactive iodine therapy, molecular imaging and serum biomarkers for differentiated thyroid cancer: 2017 guidelines of the French Societies of Nuclear Medicine, Endocrinology, Pathology, Biology, Endocrine Surgery and Head and Neck Surgery. Ann Endocrinol (Paris). 2017 Jul;78(3):162-175. doi: 10.1016/j.ando.2017.04.023. Epub 2017 Jun 1. No abstract available. PMID 28578852
- [Background] Nixon IJ, Whitcher MM, Palmer FL, Tuttle RM, Shaha AR, Shah JP, Patel SG, Ganly I. The impact of distant metastases at presentation on prognosis in patients with differentiated carcinoma of the thyroid gland. Thyroid. 2012 Sep;22(9):884-9. doi: 10.1089/thy.2011.0535. Epub 2012 Jul 24. PMID 22827579
- [Background] de la Fouchardiere C, Alghuzlan A, Bardet S, Borget I, Borson Chazot F, Do Cao C, Godbert Y, Leenhardt L, Zerdoud S, Leboulleux S. The medical treatment of radioiodine-refractory differentiated thyroid cancers in 2019. A TUTHYREF(R) network review. Bull Cancer. 2019 Sep;106(9):812-819. doi: 10.1016/j.bulcan.2019.04.012. Epub 2019 Jun 11. PMID 31200896
- [Background] Schlumberger M, Tahara M, Wirth LJ. Lenvatinib in radioiodine-refractory thyroid cancer. N Engl J Med. 2015 May 7;372(19):1868. doi: 10.1056/NEJMc1503150. No abstract available. PMID 25946295
- [Background] Fugazzola L, Elisei R, Fuhrer D, Jarzab B, Leboulleux S, Newbold K, Smit J. 2019 European Thyroid Association Guidelines for the Treatment and Follow-Up of Advanced Radioiodine-Refractory Thyroid Cancer. Eur Thyroid J. 2019 Oct;8(5):227-245. doi: 10.1159/000502229. Epub 2019 Aug 28. PMID 31768334
- [Background] Durante C, Haddy N, Baudin E, Leboulleux S, Hartl D, Travagli JP, Caillou B, Ricard M, Lumbroso JD, De Vathaire F, Schlumberger M. Long-term outcome of 444 patients with distant metastases from papillary and follicular thyroid carcinoma: benefits and limits of radioiodine therapy. J Clin Endocrinol Metab. 2006 Aug;91(8):2892-9. doi: 10.1210/jc.2005-2838. Epub 2006 May 9. PMID 16684830
- [Background] Keutgen XM, Sadowski SM, Kebebew E. Management of anaplastic thyroid cancer. Gland Surg. 2015 Feb;4(1):44-51. doi: 10.3978/j.issn.2227-684X.2014.12.02. PMID 25713779
- [Background] Ibrahimpasic T, Ghossein R, Shah JP, Ganly I. Poorly Differentiated Carcinoma of the Thyroid Gland: Current Status and Future Prospects. Thyroid. 2019 Mar;29(3):311-321. doi: 10.1089/thy.2018.0509. PMID 30747050
- [Background] Lazar V, Bidart JM, Caillou B, Mahe C, Lacroix L, Filetti S, Schlumberger M. Expression of the Na+/I- symporter gene in human thyroid tumors: a comparison study with other thyroid-specific genes. J Clin Endocrinol Metab. 1999 Sep;84(9):3228-34. doi: 10.1210/jcem.84.9.5996. PMID 10487692